CLINICAL TRIAL: NCT04401254
Title: The Coronavirus Disease 2019 - Recovery Study
Brief Title: Recovery of Patients From COVID-19 After Critical Illness
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-Recovery V1.5 9Feb2022
Record Dates: First submitted 2020-05-07; First posted 2020-05-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; Critical Illness
Keywords: recovery
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who are critically ill with COVID-19 requiring life support in an intensive care unit (ICU) have increased risk of morbidity and mortality. Currently the ICU community does not know what effect the disease, the ICU admission, physiotherapy interventions and life support have on their long-term quality of life and whether they can return to their pre-illness level of function following ICU.

COVID-Recovery will describe the physiotherapy interventions delivered to critically ill patients with COVID-19. In survivors, COVID-Recovery will utilise telephone follow-up of ICU survivors to assess disability-free survival and quality of life at 6 months after ICU admission. Additionally, COVID-Recovery will identify if there are predictors of disability-free survival. COVID-Recovery will aim to select up to 300 patients diagnosed with COVID-19 from ICUs in Australia. If they survive to hospital discharge, patients will be invited to receive a telephone questionnaire at 6 months after the ICU admission that aims to assess their long-term outcomes, including physical, cognitive and emotional function, quality of life, and whether they have been able to return to work following ICU discharge.

To describe the experience of critical illness in survivors of COVID-19 and their family members.

To explore and describe functional recovery, respiratory system function and respiratory health morbidity up to 6 months after ICU admission in persistently critically ill adults with COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19 patients who have been admitted to ICU for > 24 hours
2. Patients aged over 17 years

Persistent critical illness cohort

1. As above
2. An ICU admission of at least 10 consecutive days

Exclusion Criteria:

* Previous enrolment in this study in a prior ICU admission

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients with COVID-19 admitted to an intensive care unit
Sampling Method: Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Disability-free survival | 6 months
  a composite measure of WHODAS 2.0 - 12 level and hospital survival
Physiotherapy intervention | During the ICU stay until 3 months
  The physiotherapy interventions provided to patients with COVID-19 admitted to the ICU and health outcomes

SECONDARY OUTCOMES:
Health status | 6 months
  Health related quality of life measured with EQ5D-5L score from 0 to 100
Global function | 6 months
  World Health Organization Disability Assessment Schedule 2.0 12L
Cognitive function | 6 months
  Montreal Cognitive Assessment Blind
Anxiety and depression | 6 months
  Hospital Anxiety and Depression Scale
Screening for post-traumatic distress | 6 months
  Impact of Events Scale Revised
Work Status | 6 months
  WHODAS 2.0
Proportion of patients with COVID-19 who received physiotherapy in ICU | During the ICU stay until 28 days
The reported barriers to delivering physiotherapy interventions | During the ICU stay until 28 days
  Physiotherapist reported barriers to delivering the intervention
Adverse events during physiotherapy interventions | During the ICU stay until 28 days
  Adverse events that require the intervention to be ceased for medical intervention
Phenomenological data of the patient and family experience | 6 months
  Qualitative interviews
Global function | 6 months
  Global Rating of Change

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, PhD, Principal Investigator — Monash University
Locations (29):
- Australia (29):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Hospital, Concord, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston Hospital, Launceston, Tasmania
  - Casey Hospital, Berwick, Victoria
  - Box Hill Hospital (Eastern Health), Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Cabrini Health, Malvern, Victoria
  - Australian New Zealand Intensive Care Research Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sunshine Hospital, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared if approved by the steering committee and with ethical approvals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after completion of the study for 12 months
Access Criteria: Email the Chief Investigator

REFERENCES:
- [Derived] Hodgson CL, Higgins AM, Bailey MJ, Mather AM, Beach L, Bellomo R, Bissett B, Boden IJ, Bradley S, Burrell A, Cooper DJ, Fulcher BJ, Haines KJ, Hodgson IT, Hopkins J, Jones AYM, Lane S, Lawrence D, van der Lee L, Liacos J, Linke NJ, Gomes LM, Nickels M, Ntoumenopoulos G, Myles PS, Patman S, Paton M, Pound G, Rai S, Rix A, Rollinson TC, Tipping CJ, Thomas P, Trapani T, Udy AA, Whitehead C, Anderson S, Neto AS; COVID-Recovery Study Investigators and the ANZICS Clinical Trials Group. Comparison of 6-Month Outcomes of Survivors of COVID-19 versus Non-COVID-19 Critical Illness. Am J Respir Crit Care Med. 2022 May 15;205(10):1159-1168. doi: 10.1164/rccm.202110-2335OC. PMID 35258437
- [Derived] Hodgson CL, Higgins AM, Bailey MJ, Mather AM, Beach L, Bellomo R, Bissett B, Boden IJ, Bradley S, Burrell A, Cooper DJ, Fulcher BJ, Haines KJ, Hopkins J, Jones AYM, Lane S, Lawrence D, van der Lee L, Liacos J, Linke NJ, Gomes LM, Nickels M, Ntoumenopoulos G, Myles PS, Patman S, Paton M, Pound G, Rai S, Rix A, Rollinson TC, Sivasuthan J, Tipping CJ, Thomas P, Trapani T, Udy AA, Whitehead C, Hodgson IT, Anderson S, Neto AS; COVID-Recovery Study Investigators and the ANZICS Clinical Trials Group. The impact of COVID-19 critical illness on new disability, functional outcomes and return to work at 6 months: a prospective cohort study. Crit Care. 2021 Nov 8;25(1):382. doi: 10.1186/s13054-021-03794-0. PMID 34749756